CLINICAL TRIAL: NCT06788522
Title: The Effects of Orexin Antagonism on Fear Extinction in PTSD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MHBP-006-24S
Record Dates: First submitted 2025-01-16; First posted 2025-01-23 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Insomnia; PTSD
Keywords: Fear conditioning; PTSD; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Stress Disorders, Post-Traumatic | interventions — suvorexant

STUDY DESIGN:
Intervention Model Description: In line with the CSRD Combined Proof of Concept and Clinical Merit Review Award mechanism, this proposal aims to conduct a proof-of-concept study that will lead to a larger clinical trial to further the evidence base for the intervention. For this study, the investigators propose a home-based multi-day remote fear conditioning experiment where nightly doses of suvorexant or placebo will be administered following extinction training over the subsequent 6 nights. In phase 1, the investigators will demonstrate our remote fear conditioning task and assess its feasibility by conducting a pilot study in which the investigators will enroll and randomize 40 Veterans with PTSD and insomnia. The design for Phase 1 (and Phase 2) will involve a double-blind, randomized, placebo-controlled experiment of suvorexant on fear extinction in a home-based classical aversive conditioning paradigm in male and female Veterans with PTSD and insomnia.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be blindly assigned to treatment according to a randomization schedule generated by the study biostatistician using a computerized allocation schedule system. Study investigators, staff, and participants will remain blinded to treatment allocation throughout the study. A study physician will prescribe the study drug and will remain blind to treatment assignment for the study duration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Suvorexant (Experimental): Suvorexant pills (10-20 mg)
  Interventions: Drug: Suvorexant
- Placebo (Placebo Comparator): Matching placebo pills
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Suvorexant — Suvorexant pills (10-20 mg)
  Arms: Suvorexant
Drug: Placebo — Matching placebo pills
  Arms: Placebo

SUMMARY:
PTSD affects approximately 22% of Veterans who have served in Iraq and Afghanistan. Symptoms of PTSD may include re-experiencing, avoidance of trauma reminders, negative thoughts or feelings, and hyperarousal, such as increased startle reactivity and disturbed sleep. Treatments for PTSD are based on fear extinction principles in which individuals are repeatedly exposed a feared cue in the absence of danger, resulting in diminishing physiological reactions, a process believed to underlie recovery from PTSD. Studies suggest that orexin, a wake-promoting neuropeptide, may enhance fear extinction. This study will examine whether suvorexant, a selective orexin-receptor antagonist, will enhance fear extinction in Veterans with PTSD and insomnia. Finding a role for orexins in fear extinction will support the rationale for its further evaluation in the treatment of PTSD. Suvorexant is an accessible, safe medication that has been well-established in treating insomnia. It has outstanding promise for treating common and distressing symptoms in Veterans with PTSD.

DETAILED DESCRIPTION:
PTSD is a common consequence of combat manifested in part by trauma-related arousal and reactivity, seen in increased startle and impaired sleep that result from central and autonomic nervous system alterations. Impaired fear extinction may explain prolonged physiological alterations in PTSD. Preclinical evidence suggests that orexin, a wake-promoting neuropeptide, may be a shared mechanism underlying both sleep and fear extinction. While rodent studies have shown that pharmacological manipulations that block orexin in rodents facilitate fear extinction, no studies have tested this in humans with PTSD.

In line with the CSRD Combined Proof of Concept and Clinical Trial Merit Review Award mechanism, the investigators propose a proof-of-concept study leading to a clinical trial. During the initial phase, the investigators will develop and establish feasibility of the task and recruitment in 40 eligible participants with PTSD and insomnia. The task will involve a home-based multi-day remote fear conditioning experimental study, in which Veterans with PTSD and insomnia will receive nightly doses of suvorexant or placebo following extinction training over the subsequent 6 nights. Primary Aims of the proof of concept will be to: 1) establish remote fear conditioning procedures collaboratively with Veteran stakeholders; 2) evaluate enrollment, tolerability, adherence, and retention; 3) demonstrate fear conditioning and extinction learning using remote procedures; and 4) determine task feasibility of the home-based remote fear conditioning task. Go/No go milestones include: 1) the ability to enroll and randomize 40 participants by the end of month 23; 2) most participants (> 80%) will take medication as prescribed over 7 nights; 3) no SAEs during the course of treatment as determined by the data monitoring committee review (DMC); 4) < 10% of post-randomization participants will drop out (<4 participants), resulting in 36 individuals who complete all study procedures by month 23; 5) successful demonstration of measurement of fear conditioning (greater skin conductance (SC) responses to CS+ cues vs CS- cues) and fear extinction (differential SC responses to CS+ and CS- cues that diminish over trials) in the combined sample; 6) feasibility of the remote task demonstrated by <15% data loss due to recording issues (e.g., technical malfunction or UCS non-response in <6 participants).

If milestones are met, the investigators will advance to a clinical mechanistic trial to evaluate suvorexant in facilitating fear extinction using a double-blind randomized, placebo-controlled experimental design in Veterans with PTSD and insomnia. A total of 120 male and female Veterans with PTSD and insomnia will be randomized to either the suvorexant or placebo condition (n=60 in each condition). Participants will be trained in multi-day remote procedures involving fear conditioning (Day 1) and extinction 3 days later (Day 4), followed by 10 mg. suvorexant or placebo. A flexible dose titration of suvorexant (10-20 mg.) or matching placebo will be administered over the next 6 nights. Participants will then undergo extinction retention and fear reinstatement tests one week after extinction (Day 11). Primary outcome measures will be differential skin conductance responses to CS+ and CS- cues during extinction retention and reinstatement phases.

Primary Aims of the Clinical Trial will be: 1) To examine whether suvorexant facilitates fear extinction, seen as greater extinction retention compared to placebo. 2) To examine whether the facilitative effects of suvorexant are more resistant to reinstatement compared to placebo. Pending an effect of suvorexant on fear extinction retention and reinstatement, the investigators will evaluate whether improvement in insomnia mediates these effects. In-home sleep recording (including both sleep EEG and indices of sleep-disordered breathing) and sleep diary measures will be examined as secondary mediators. Greater improvement in sleep quality will partially account for greater extinction retention and less reinstatement. If successful, the proposed study will offer proof-of-concept data and meaningful guidance for future studies of suvorexant as an augmentation co-treatment in exposure therapy.

ELIGIBILITY:
Inclusion Criteria:

* (same for Phase 1 and Phase 2):

  * men and women
  * a history of US military service
  * capable of reading and understanding English
  * able to provide written informed consent
* Criterion A event meets DSM-5 criteria and occurred during military service, including combat and military sexual trauma
* Chronic full PTSD diagnosis >3 months duration as indexed by CAPS-5 at screening, and CAPS-5 score > 30
* Insomnia indicated by insomnia severity index (ISI) score > 14
* Subjects on non-exclusionary medications, and must be on a stable dose for at least 4 weeks prior to randomization, including Selective Serotonin Reuptake Inhibitors (SSRIs, e.g.,):

  * sertraline
  * paroxetine
  * fluoxetine
  * fluvoxamine
  * citalopram
  * escitalopram
* Serotonin-norepinephrine reuptake inhibitors (SNRIs; e.g.):

  * Desvenlafaxine
  * Duloxetine
  * Levomilnacipran
  * Venlafaxine
* For subjects who are in psychotherapy, treatment must be stable for 6 weeks
* Women of child-bearing potential must not be pregnant or have plans for pregnancy or breastfeeding during the study and must use a medically acceptable method of birth control

Exclusion Criteria:

* Moderate or severe DSM-5 alcohol or cannabis use disorder in the last 3 months

  * Mild alcohol use disorder with abstinence of 30 days will be allowed
  * Mild marijuana use disorder will be allowed with abstinence for one week prior to participation
  * Any other DSM-5 drug use disorder in the last 3 months will be excluded
* Lifetime bipolar disorder I or II, schizophrenia, schizoaffective disorder, obsessive-compulsive disorder, or major depressive disorder with psychotic features
* Exposure to trauma in the last 3 months
* Use of exclusionary antidepressant (trazodone, mirtazapine, doxepin, tricyclics), mood stabilizers (e.g., lithium), antipsychotic medication
* Prominent suicidal or homicidal ideation or any suicidal behavior in the past 3 months on the Columbia Suicide Severity Rating Scale (C-SSRS) or increased risk of suicide that necessitates additional therapy or inpatient treatment
* Pre-existing moderate sleep apnea or positive screen for sleep apnea by type III device (AHI>15) in the absence of adherence to effective treatment (such as CPAP or oral device)
* Night shift work or extreme morning or evening tendencies in order to avoid the impact of circadian factors on subjective and objective sleep measures
* Neurologic disorder or systemic illness affecting CNS function
* Chronic or unstable medical illness, including:

  * unstable angina
  * myocardial infarction within the past 6 months
  * congestive heart failure
  * preexisting hypotension or orthostatic hypotension
  * heart block or arrhythmia
  * chronic renal or hepatic failure
  * pancreatitis
  * severe chronic obstructive pulmonary disease
* History of severe traumatic brain injury as assessed by the Ohio State University Traumatic Brain Injury Identification Method (OSU-TBI ID)
* Uncorrected hearing impairment
* Mild cognitive impairment assessed by the Montreal Cognitive Assessment (MOCA)
* Pregnancy, breastfeeding and/or refusal to use effective birth control (for women)
* Previous adverse reaction to a hypnotic
* Current use of benzodiazepines, strong inhibitors of CYP3A, or Digoxin

  * The investigators will require that all participants do not consume heavy amounts of alcohol per week (>7 drinks for women, >14 drinks for men) or use illicit drugs for one week prior to participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40120 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2032-03-01 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
enrollment | Month 4-23
  Goal of enrolling 40 individuals to achieve a total of 30 completers by the end of month 23.
Medication Adherence | Month 4-23
  Pill count and adherence to instructions over 7 study nights
side effect reports | Month 4-23
  SAEs
Post-randomization drop out | Month 4-23
  Post-randomization drop-out rates
Fear conditioning and extinction | Month 4-23
  Fear conditioning (greater SC responses to CS+ cues vs CS- cues) and fear extinction (differential SC responses to CS+ and CS- cues that diminish over repeated trials) in the combined sample
Rates of technical malfunction | Month 4-23
  Rates of technical malfunction (SC levels that are missing or <.02 microsiemens) and or non-responding to the UCS (e.g., SCR<.05 microsiemens)
Electrodermal Activity | Years 2-7
  Differential SC responses to CS+ and CS- cues during extinction retention and 2) during reinstatement.

SECONDARY OUTCOMES:
Insomnia Severity Index | Years 2-7
  Self-reported sleep
Sleep EEG | Years 2-7
  Total sleep time, REM

CONTACTS AND LOCATIONS:
Overall Officials: Sabra S Inslicht, PhD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (2):
- United States (2):
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No